CLINICAL TRIAL: NCT00857974
Title: Impact of a Physical Activity Intervention on Physical Function and Quality of Life in Aging Candidates for Renal Transplantation: The PART Study
Brief Title: Physical Activity Program for Older Renal Transplant Candidates
Acronym: PART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: The John A. Hartford Foundation (Other); Association of Subspecialty Professors (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001451
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Renal Transplant Candidate
Keywords: Physical Activity; Renal Transplant Candidate; Physical Function; Body Composition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): No physical activity intervention will be prescribed for the Usual Care Arm.
- Physical Activity (Active Comparator)
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Physical Activity — The intervention is an individualized, structured, moderate intensity home-based physical activity program. During the first 12 weeks the program will focus on lower extremity strengthening, and thereafter incorporate cardiovascular activity. The target duration of activity is 150 minutes per week, i.e., 20-30 min on most days of the week. However, the program is adjusted based on each participant's progression, initial level of physical fitness and will be modified in response to illness, injury, or physical symptoms.
  Arms: Physical Activity

SUMMARY:
The physical function of older candidates for renal transplantation and their ability to sustain physical activity programs are currently unknown. The primary goal of this study is to determine the feasibility of a physical activity intervention in older dialysis-dependent patients, assessing its effect on maintaining transplant candidacy and outcome after transplantation. Clinical practice guidelines do not set an absolute age limit for evaluating potential renal transplant candidates. While cardiovascular risk assessment and malignancy screening are emphasized in the older age group, physical performance and the risk for disability are often overlooked. Although healthy older patients experience increased life expectancy after renal transplantation versus remaining on dialysis, outcomes such as the capacity to live independently and function well have not been studied. Given the poorer baseline health status in aging end-stage renal disease patients, rapid changes in health on dialysis, and the national organ shortage, it is increasingly important to identify factors that predict better outcomes and devise strategies that will maximize the benefit of transplantation in older individuals.

The investigators hypothesize that muscle is the principal organ system underlying impaired physical function among older transplant candidates, and that decreased muscle mass and physical functioning lead to poorer outcomes in older renal transplant candidates. The investigators propose that a simple bedside performance measurement of lower extremity functional limitations, the Short Physical Performance Battery, will be a strong predictor of outcomes in this patient cohort. The investigators also propose that outcomes can be improved with exercise training, potentially leading to longer durations of active transplant candidacy and greater independence after successful transplantation. The Specific Aims of this research are:

1. Determine the feasibility of an exercise intervention in dialysis-dependent wait-listed patients age 60 years and over who will be randomized to one of two groups: usual care versus a structured physical activity program.
2. Define the natural history of physical function in patients age 60 years and greater who remain on dialysis or undergo renal transplantation attempting to identify a subgroup of older wait listed patients who are at high risk for developing disability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Listed on the renal transplant waiting list (either active or inactive status)
* Able to give consent
* Able to maintain sitting or standing balance and ambulate without assistance from another person

Exclusion Criteria:

* MMSE score less than 21
* Unstable coronary artery disease
* Less than three months since the patient had a myocardial infarction
* Congestive heart failure NY class III or IV
* Lower extremity amputation without prosthesis
* Severe and active lower extremity musculoskeletal problem which prevents participation in the intervention
* Individuals who are more active than the intervention and thus would not be likely to benefit
* SPPB score of 12 (the maximum score) at screening

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The Short Physical Performance Battery SPPB) score, a brief and simple bedside performance-based instrument. | One year

SECONDARY OUTCOMES:
Health-related quality-of-life scores | One year
Self-reported disability scores | One year
Re-hospitalization | One year
Inter-current illness including cardiovascular events or falls | One year
Endurance | One year
Body composition by both DEXA and thigh CT | One year
Grip strength | One year
Leg strength | One year
ADL disability | One year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kritchevsky, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States